CLINICAL TRIAL: NCT01812382
Title: A Study to Evaluate the Feasibility of Microdialysis to Determine Skin Concentrations of Retapamulin in Healthy Volunteers
Brief Title: Retapamulin Microdialysis Feasibility Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117151
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Skin Infections, Bacterial
Keywords: Penetration; Antibiotic; Microdialysis; Formulation Pharmacokinetics; Feasibility
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Microdialysis arm (Experimental): Three microdialysis probes will be placed in the thigh of each subject prior to the start of the microdialysis procedure/infusion using a microdialysis device. All subjects will receive Sodium Chloride solution perfused for 30 minutes followed by Retapamulin perfusion for 90 minutes and then Saline perfusion will occur during the washout period.
  Interventions: Drug: Retapamulin Microdialysis

INTERVENTIONS:
Drug: Retapamulin Microdialysis — After a 30 minutes equilibration period of the microdialysis procedure/infusion with normal saline solution, 50nanogram (ng)/mL Retapamulin injectable solution will be infused at a flow rate of 1.5 microliter/minute over a period of 90 minutes. The total dose perfused for each of the 3 microdialysis tubes will be 6.75ng.

SUMMARY:
This feasibility study will allow for the determination of the in vivo recovery and time of dialysis to optimize a future thorough microdialysis study. This is a single session, open label study to evaluate the feasibility of microdialysis for Retapamulin in healthy subjects. Three healthy subjects will be enrolled and complete the study procedures. Subjects will be admitted to the research unit on Day 1 and three microdialysis probes will be placed in the thigh of each subject prior to the start of the microdialysis procedure. After normal saline solution infusion for 30 minutes, a Retapamulin solution will be infused for 90 minutes. Saline perfusion will occur during the washout period. Microdialysis sampling will be done for 30 minutes (during the last 30 minutes of drug perfusion) and dialysate sample collection will continue every 30 minutes for 4 hours. The approximate duration of study including follow-up is 4 days.

ELIGIBILITY:
Inclusion Criteria:

Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with clinically significant lab values outside the normal range should always be excluded from enrollment.

* The subject is able to understand and comply with protocol requirements, instructions and protocol-stated restrictions and is likely to complete the study as planned. Subject is willing to provide informed consent.
* Does not use medications containing Retapamulin while participating in the study.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* Body Mass Index within the range 18.5 to 32 kilogram/ meter^2 (inclusive).
* The following normal ranges for blood pressure and heart rate are given as a guide: Systolic blood pressure 90 to 140 milimeter of Mercury (mmHg), Diastolic blood pressure 60 to 90 mmHg, and Heart rate 45 to 100 beats per minute (bpm). The investigator may interpret screening vital sign data based on the subject's age, physical state and level of fitness. Subjects with vital sign readings marginally outside the normal range may be included in the study if in the investigator's opinion these values are not clinically significant and will not present a safety risk or affect study assessments.
* A female subject is eligible to participate if she is of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone > 40 milli international unit/mililiter (mL) and estradiol < 40 picogram/ml [<147 picomoles/Liter] is confirmatory]. Females on hormone replacement therapy and whose menopausal status is in doubt will be required to use one of the contraception methods) or Child-bearing potential and agrees to use one of the contraception methods for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until study completion (i.e. follow-up phone call). Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until study completion (i.e. follow-up phone call).
* Alanine aminotransferase, alkaline phosphatase and bilirubin <= 1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* QT interval corrected for Heart rate (QTc), QTcB (Bazett's formula) or QTcF (Fridericia's formula) < 450 millisecond (msec); or QTc < 480 msec in subjects with Bundle Branch Block.
* Does not currently smoke cigarettes or tobacco and has not smoked within the past 12 months prior to the study.
* Does not consume alcohol 72 hours prior to the start of and during the study

Exclusion Criteria:

* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated.
* History of current significant medical illness including cardiovascular thrombotic events, myocardial infarction, stroke or other cardiac disease, hypertension, peptic ulcer disease or gastrointestinal bleeding, skin disorders, hematological disease, bronchospastic respiratory disease, asthma, diabetes mellitus, renal or hepatic insufficiency, or any other illness that the investigator deems clinically significant for exclusion of the subject from the study.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of skin conditions including atopic dermatitis, dry skin, or ichtyosis vulgaris.
* Surgical history within 3 months prior to the start of the study.
* Clinically significant acute illness 7 days prior to study start.
* Excessive hair, tattooing, scar tissue, or other tissue damage at the application site that could affect drug recovery or patient safety.
* Use of topical moisturizers (does not include facial moisturizers) 48 hours before the start of and during the study.
* Strenuous exercise 48 hours before the start of and during the study.
* Unable to refrain from the use of non-prescription drugs, including non- steroidal ant-inflammatory drugs (NSAIDS), vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360mL) of beer; 5 ounces (150mL) of wine; or 1.5 ounce (45mL) of 80 proof distilled spirits.
* A positive pre-study drug/alcohol screen.
* Pregnant females as determined by positive serum human chorionic gonadotropin (hCG) at screening or urine hCG test prior to dosing.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Employees of the investigator or study center, with direct involvement in the proposed study or similar studies including family members of the employees or the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2014-05-27 (Actual); Study Completion 2014-05-27 (Actual)

PRIMARY OUTCOMES:
Retapamulin concentrations in the dialysate samples | Single day
  Retapamulin concentrations in the dialysate samples will be collected to calculate the length of time needed until disappearance of the drug in the dialysate (washout) and the percentage of drug recovered following perfusion of Retapamulin solution by microdialysis to the thigh of healthy volunteers. Microdialysis is a minimally-invasive sampling technique that is used for continuous measurement of free, unbound analyte concentrations in the extracellular fluid of virtually any tissue

SECONDARY OUTCOMES:
Safety and tolerability of the microdialysis technique with perfused Retapamulin assessed by number of participants with Adverse Events (AEs) | Up to 4 days
  Adverse event collection and recording will begin with first dose and continue until the final follow-up visit
Safety and tolerability of the microdialysis technique with perfused Retapamulin assessed by Laboratory parameters | Single day
  Laboratory parameters include: Hematology, Clinical Chemistry and additional parameters
Safety and tolerability of the microdialysis technique with perfused Retapamulin assessed by Vital Sign measurements | Single day (Pre-dose and at 7th hour Post-dose)
  Vital Signs include: Systolic and Diastolic Blood Pressure and Pulse Rate. Pre-dose Vital Signs will be performed in triplicate and all other will be done in duplicate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 117151 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/117151?search=study&search_terms=117151#rs
- Available data/document: Dataset Specification: 117151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117151 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register